CLINICAL TRIAL: NCT00196924
Title: Evaluate the Safety and Immunogenicity of GSK Biologicals' HPV-16/18 Vaccine Administered Intramuscularly According to a 0,1,6 Month Schedule in Healthy Female Subjects (10 - 14 Years)
Brief Title: Human Papilloma Virus Vaccine Safety and Immunogenicity Trial in Young Adolescent Women With GSK Bio HPV-16/18.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 580299/013
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: HPV-16/18 L1/AS04

SUMMARY:
Human Papilloma virus (HPV) are viruses that cause a common infection of the skin and genitals in men and women. Several types of HPV infection are transmitted by sexual activity and, in women, can infect the cervix (part of the uterus or womb). This infection often goes away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. If a woman is not infected by HPV, it is very unlikely that she will get cervical cancer. This study will evaluate the safety and immunogenicity of GSK Biologicals HPV-16/18 vaccine over 12 months, in pre-teen and adolescent women of 10-14 years of age at study start. Approximately 2000 study subjects will receive the HPV vaccine or a control vaccine (hepatitis A vaccine) administered intramuscularly according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria:

A woman between, and including, 10 and 14 years of age at the time of the first vaccination.

Written informed consent from the subject prior to enrolment. Subject must be free of obvious health problems. Subject must have negative urine pregnancy test.

Exclusion Criteria:

Pregnant or breastfeeding. Known acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality.

History of chronic condition(s) requiring treatment such as cancer, chronic hepatitis or kidney disease(s), diabetes, or autoimmune disease.

Previous vaccination against human papillomavirus (HPV).

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2067 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Demonstration of safety of the HPV vaccine compared to the control (occurrence of SAEs) up to month 7.

SECONDARY OUTCOMES:
Safety of HPV vaccine in entire study period. Vaccine immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (55):
- Australia (2):
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Perth, Western Australia
- GSK Investigational Site, Bogotá, Colombia
- Czechia (2):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Pardubice
- France (11):
  - GSK Investigational Site, Aubevoye
  - GSK Investigational Site, Broglie
  - GSK Investigational Site, Évreux
  - GSK Investigational Site, Luynes
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nogent-le-Roi
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pont-de-l'Arche
  - GSK Investigational Site, Saint-Sébastien-de-Morsent
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Verneuil-sur-Avre
- Germany (23):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bützow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Brunsbüttel, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Harrislee, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Niebüll, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Weimar, Thuringia
- GSK Investigational Site, Comayagüela, Honduras
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
- GSK Investigational Site, Ciudad de Panama - La Chorrera, Panama
- GSK Investigational Site, Seoul, South Korea
- Spain (6):
  - GSK Investigational Site, Alcora/Castellón
  - GSK Investigational Site, Alquerías Del Niño Perdido (Castellón)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Örebro
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tao Yuan County

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Boxus M, Lockman L, Fochesato M, Lorin C, Thomas F, Giannini SL. Antibody avidity measurements in recipients of Cervarix vaccine following a two-dose schedule or a three-dose schedule. Vaccine. 2014 May 30;32(26):3232-6. doi: 10.1016/j.vaccine.2014.04.005. Epub 2014 Apr 13. PMID 24731816
- [Derived] Schwarz TF, Huang LM, Medina DM, Valencia A, Lin TY, Behre U, Catteau G, Thomas F, Descamps D. Four-year follow-up of the immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine when administered to adolescent girls aged 10-14 years. J Adolesc Health. 2012 Feb;50(2):187-94. doi: 10.1016/j.jadohealth.2011.11.004. PMID 22265115
- [Derived] Medina DM, Valencia A, de Velasquez A, Huang LM, Prymula R, Garcia-Sicilia J, Rombo L, David MP, Descamps D, Hardt K, Dubin G; HPV-013 Study Group. Safety and immunogenicity of the HPV-16/18 AS04-adjuvanted vaccine: a randomized, controlled trial in adolescent girls. J Adolesc Health. 2010 May;46(5):414-21. doi: 10.1016/j.jadohealth.2010.02.006. PMID 20413076
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 580299/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 580299/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 580299/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 580299/013 are summarised with studies 104896 (M18), 104902 (M24), 104904 (M36) and 104918 (M48) on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 580299/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 580299/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 580299/013 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register